CLINICAL TRIAL: NCT07192562
Title: The Effects of Virtual Reality-Based Exercise Games on Physical and Cognitive Health in Sedentary Workplace Employees
Brief Title: Effects of VR-Based Exergames on Physical and Cognitive Health in Sedentary Workers
Acronym: VR-Exergame
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Hakan GÜLER, MSc, Audiologist, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HGULER; BAP-2024/57 No:E-93425710-604 (Other Grant/Funding Number: Medipol University, Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2025-09-09; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Virtual Reality Therapy
Keywords: Sedentary Lifestyle; Virtual Reality Exercise; Exergames; Balance; Cognitive Function
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: This was a two-arm, parallel-group, randomized controlled trial. Participants were randomly assigned in a 1:1 ratio to either the VR Exercise Group or the Control Group. The VR group received a 6-week virtual reality-based exercise intervention (two sessions per week, ~30-35 minutes each), while the Control group continued their usual daily routines without structured exercise.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments were performed by evaluators who were blinded to group allocation, ensuring a single-blinded study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Exercise Group (Experimental): Participants performed a virtual reality-based exercise program using the Meta Quest 2 headset. Two commercial exergames (Beat Saber and PowerBeatsVR) were implemented twice weekly for six weeks (12 sessions total). Each session lasted approximately 30-35 minutes and included full-body movements such as punching, squatting, dodging, and stepping.
  Interventions: Behavioral: Virtual Reality-Based Exercise Program
- Control Group (No Intervention): Participants did not receive any structured exercise intervention and continued their usual daily routines throughout the 6-week study period.

INTERVENTIONS:
Behavioral: Virtual Reality-Based Exercise Program — Participants in the VR Exercise Group received a virtual reality-based physical activity intervention using the "Meta Quest 2" headset. Two exergames, "Beat Saber" and "PowerBeatsVR", were implemented twice a week for six weeks, totalling 12 exercise sessions. Each session lasted 30-35 minutes and was conducted individually during work hours. Beat Saber provided rhythm-based tasks involving block slicing and obstacle dodging, while PowerBeatsVR included high-intensity punching, squatting, and side-stepping movements. Game difficulty increased weekly.
  Arms: Virtual Reality Exercise Group

SUMMARY:
Sedentary behavior in the workplace is associated with declines in both physical and cognitive health. Traditional exercise programs are often difficult to sustain among workplace employees, leading to an increased interest in digital and interactive solutions such as virtual reality (VR)-based exergames.

This randomized controlled study investigated the feasibility and effects of a VR-based exercise intervention on physical and cognitive outcomes in sedentary university employees. A total of 32 participants aged 30-60 years with low physical activity levels (<600 MET-min/week) were recruited and randomized into two groups: VR Exercise (n=16) and Control (n=16).

Participants in the VR Exercise Group received a virtual reality-based physical activity intervention using the "Meta Quest 2" headset. Two exergames, "Beat Saber" and "PowerBeatsVR", were implemented twice a week for six weeks, totalling 12 exercise sessions. Each session lasted 30-35 minutes and was conducted individually during work hours. Beat Saber provided rhythm-based tasks involving block slicing and obstacle dodging, while PowerBeatsVR included high-intensity punching, squatting, and side-stepping movements.Game difficulty increased weekly (Figure 2). Adverse events (eg, cybersickness, dizziness, nausea) were monitored throughout each session. No adverse events were reported in either group. According to the Virtual Reality Institute of Health and Exercise, Beat Saber is classified as a moderate-intensity activity, while PowerBeatsVR is classified as high-intensity , which supports the game selection rationale in this study. Participants' sessions were monitored using a Huawei D15 laptop, and a safety boundary was configured using the VR system's room-scale feature.

Balance was assessed using the Becure Balance System and Flamingo Balance Test, while cognitive performance was measured with the CNS Vital Signs battery, which evaluates domains such as memory, attention, processing speed, and executive function. BMI was also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Being between 30-60 years of age

Being employed as an academic or administrative employees member at a university

Classified as inactive (sedentary) according to the International Physical Activity Questionnaire-Short Form (IPAQ-SF) results

Not starting any regular physical activity programs during the study period

Having normal blood pressure and circulatory conditions

No conditions preventing the use of VR technology and games (e.g., severe motion sickness)

Voluntarily agreeing to participate in the study and providing written informed consent

Exclusion Criteria:

* Pregnancy

Presence of neurological and/or psychological disorders

Having cardiovascular, respiratory, joint, or other orthopedic conditions that would prevent safe participation in exercise

Presence of vestibular disorders

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Postural Balance Performance | Baseline and 6 weeks post-intervention
  Postural balance was objectively measured using the Becure Balance System, a low-cost, portable force platform enhanced with sensors. Six sub-tests were conducted: double-leg stance with eyes open/closed, single-leg stance (right/left), foam surface double-leg stance with eyes open/closed. The system provides real-time feedback and detailed reports on postural sway and center of pressure (COP) movement .
Cognitive Performance | Baseline and 6 weeks post-intervention
  Cognitive functions were evaluated using the CNS Vital Signs test battery, which provides scores for domains such as psychomotor speed, processing speed, motor speed, memory, and executive function. Higher scores indicate better performance.
Body Mass Index (BMI) | Baseline and 6 weeks post-intervention
  BMI was calculated as body weight in kilograms divided by height in meters squared (kg/m²). No additional interventions for weight control were provided.
Change in Static Balance | Time Frame: Baseline and 6 weeks post-intervention
  Flamingo Balance Test: This Eurofit static balance test assessed participants' ability to maintain balance on a wooden beam (50 cm long, 5 cm high, 3 cm wide) using their dominant leg. Total loss of balance within 60 seconds was recorded. If more than 15 falls occurred in the first 30 seconds, the test was terminated and scored zero.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol Universıty, Beykoz, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared.